CLINICAL TRIAL: NCT03630965
Title: Audiovisual Tool Use in the ICU, to Impact the Anxiety Level of Patients' Surrogates While Deciding on Cardiopulmonary Resuscitation
Brief Title: CPR Audiovisual Tool to Impact ICU Patients' Surrogate Anxiety Level.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Tirsa M. Ferrer Marrero, Primary Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PULM-AV-CPR; PRO00029203 (Medical College of Wisconsin)
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): No CPR video
- Group B (Experimental): CPR video
  Interventions: Other: CPR Video

INTERVENTIONS:
Other: CPR Video — A 7.07 minutes' CPR video will be administered to the ICU patients' surrogates in Group B.
  After viewing the video, the surrogate will complete the Hamilton Anxiety Rating Scale, a five-question survey about CPR, and a one-question form about comfort using the Likert Scale.
  Arms: Group B

SUMMARY:
Video or No Video to decrease HCPOA/LAR anxiety and increase knowledge as it pertains to CPR.

DETAILED DESCRIPTION:
Designated surrogate decision makers of 30 medical intensive care unit patients will be consented and enrolled to receive either a video describing CPR and it's outcomes after standard of care code discussions versus standard of care code discussions alone. All participants will complete a short questionnaire to determine their knowledge level regarding CPR and to assess their anxiety levels. Patients who view the video will also rate their comfort level while watching the video on a 5 point Likert scale.

ELIGIBILITY:
Surrogate decision maker or power of attorney identified within the first 48 hours of ICU admission.

Surrogates or power of attorney over the age of 18 y/o

Secondary Subjects:

* Admitted to the ICU
* Critically ill to the point of treating team discussing code status with LAR/POA/Family

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Measure the impact of CPR video on the Surrogate's level of anxiety during the decision-making process on code status, in the ICU compared to the control group of surrogates (No intervention group). | 2.5 years
  30 surrogates in the ICU (15 in the intervention group and 15 in the No intervention group) will be administered the validated Hamilton Anxiety Rating Scale (HAM-A), to measure the surrogates' anxiety level . The HAM-A questionnaire has been validated to assess for anxiety, and classify anxiety.
  The Score in HAM-A is on a scale of 0 to 56 total score, when it is less than 17 there is no anxiety or mild; 18-24 is mild to moderate; 25-30 is moderate to severe; and 30-56 is severe anxiety.
  The HAM-A questionnaire has been validated to assess change in anxiety after an intervention or treatment, with a delta in total score of 8 with a Standard deviation of 1.7.

SECONDARY OUTCOMES:
Measure the impact of CPR video on patients' surrogate's knowledge about CPR, when compared to the No intervention group. | 3 years
  Knowledge assessment will be performed with a 5 questions (1 point each) questionnaire.
Analyze the surrogates' comfort when watching the video. | 3 years
  Surrogate in the intervention group will be asked if he or she if feeling comfortable watching the video. This will be a single question that will be answered using a Likert Scale.
Describe if the CPR video's impact on surrogates' anxiety level, is affected by the patient's severity of illness as per the SOFA score. | 3 years
  Will calculate patients' SOFA score which is the Sequential Organ Failure Assessment (SOFA) score. It is used to grade patients' severity of organs dysfunction and mortality. The SOFA Score is on a scale of 0-24, with higher numbers correlating with higher organs dysfunction and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Tirsa Ferrer Marrero, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin/Froedtert Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Ferrer Marrero TM, Barash M, Jaber B, Nothem M, Shah K, Weber MW, Zellner Jones S, Kennedy P, Graf J, Broaddrick S, Garacci Z, Banerjee A, Kryworuchko J, Patel J. The impact of a cardiopulmonary resuscitation video on reducing surrogates' anxiety: A pilot randomized controlled trial. J Crit Care. 2021 Apr;62:235-242. doi: 10.1016/j.jcrc.2020.11.001. Epub 2020 Dec 3. PMID 33450473